CLINICAL TRIAL: NCT06989645
Title: A Prospective, Double-blinded, Randomized, Placebo-controlled Phase 1/2a Study to Assess Safety, Tolerability, Systemic Exposure, and Preliminary Efficacy of Single Intraarticular Injections of 3 Dose Levels of SYN321 and Placebo in Patients With Symptomatic Knee Osteoarthritis
Brief Title: A Phase 1/2a Study to Evaluate Single Intraarticular Injections of 3 Dose Levels of SYN321 and Placebo in Patients With Symptomatic Knee Osteoarthritis
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Synartro AB (Industry)
Collaborators: CTC Clinical Trial Consultants AB (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Basic Science
Other Study IDs: SYN321-01; 2024-517920-21-00 (EU CTIS Number)
Record Dates: First submitted 2025-05-16; First posted 2025-05-25 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-08

CONDITIONS: Osteoarthritis of Knee
Keywords: knee osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Double blind-trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- SYN321, dose level 1 (Active Comparator): Cohort 1: 6 participants recieves SYN321.
  Interventions: Drug: SYN321
- SYN321, dose level 2 (Active Comparator): Cohort 2: 6 participants recieves SYN321.
  Interventions: Drug: SYN321
- SYN321, dose level 3 (Active Comparator): Cohort 3: 6 participants recieves SYN321.
  Interventions: Drug: SYN321
- SYN321, dose level 1,2 or 3 (Active Comparator): Cohort 4: 6 participants recieves SYN321.
  Interventions: Drug: SYN321
- Placebo (Placebo Comparator): Placebo: 2 participants each from cohort 1, 2 and 3, and 6 participants from cohort 4 receive placebo.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: SYN321 — Intra-articular
  Arms: SYN321, dose level 1; SYN321, dose level 1,2 or 3; SYN321, dose level 2; SYN321, dose level 3
Drug: Placebo — Intra-articular
  Other Names: NaCl 9 mg/mL
  Arms: Placebo

SUMMARY:
This is a, phase 1/2a trial, to assess the safety, tolerability, systemic exposure as well as preliminary efficacy following a single intra-articular injection of 3 dose levels of SYN321 in patients with symptomatic knee osteoarthritis (KOA).

DETAILED DESCRIPTION:
Participants will receive a single intra-articular injection of SYN321 or placebo. 4 sequential cohorts are planned. The fourth cohort will repeat one of the previously 3 administered dose levels. The first 2 participants in each cohort will be dosed in a sentinel fashion. The participants will be followed for 56 days.

ELIGIBILITY:
Inclusion Criteria:

1. Willing and able to give electronically informed consent for participation in the trial and willing and able to participate in all procedures and follow-up evaluations necessary to complete the trial.
2. Male or female patient clinically diagnosed with KOA, no later than 3 months prior to Visit 1. The KOA diagnosis should be confirmed in the patient's medical record.
3. Dominant pain in one knee due to KOA with weight bearing pain between 4 and 8 inclusive on the NRS scale (0-10) at the time of inclusion (checked at screening [Visit 1] and confirmed at Visit 2, pain during the last 7 days).
4. Age 40 to 79 years, inclusive at the time of Visit 1.
5. Body mass index (BMI) ≥ 18.5 and < 35.0 kg/m2.
6. Patients without abnormal clinically significant medical history, physical findings, vital signs, hypotension, cardiovascular disease, ECG, and laboratory values at the time of the screening visit, as judged by the Investigator. (Discussion is encouraged between the Investigator and the Medical Monitor regarding the clinical relevance of any abnormal laboratory value during the pre-dose period.)
7. Patient is willing to discontinue all pain medication (COX-2 inhibitors, NSAIDs, and opioid analgesics) at least 10 days before trial drug administration (prior to Day 1) and for the trial duration. Paracetamol will be allowed as rescue medication up to max 4000 mg/day (except for 24 hours prior to visit to the trial site).
8. Patient agrees not to take additional knee symptom-modifying drugs (e.g., glucosamine, collagen, HA) at least 10 days before trial drug administration (prior to Day 1) and for the trial duration.
9. WOCBP must practice abstinence heterosexual intercourse (only allowed when this is the preferred and usual lifestyle of the patient) or agree to use a highly effective method of contraception with a failure rate of < 1 % to prevent pregnancy from that least 2 weeks prior to the administration of IMP to 4 weeks after the last administration of IMP. In addition, any male partner of a female patient must, unless he has undergone vasectomy, agree to use a condom from the first administration of IMP until 4 weeks after the last administration of IMP.

   The following are considered highly effective methods of contraception:
   * combined (estrogen and progestogen containing) hormonal contraception associated with inhibition of ovulation (oral, intravaginal, transdermal),
   * progestogen-only hormonal contraception associated with inhibition of ovulation (oral, injectable, implantable),
   * intrauterine device [IUD]or intrauterine hormone-releasing system [IUS]). WOCBP must refrain from donating eggs from the first IMP administration until 3 months after the last IMP administration.

   Women of non-childbearing potential are pre-menopausal females who have undergone any of the following surgical procedures; hysterectomy, bilateral salpingectomy, or bilateral oophorectomy, or who are post-menopausal defined as 12 months of amenorrhea (in questionable cases a blood sample with detection of follicle stimulating hormone [FSH] >25 IU/L is confirmatory).

   Male patients must be willing to use condom or be vasectomized or practice sexual abstinence from heterosexual intercourse (only allowed when this is the preferred and usual lifestyle of the patient) to prevent pregnancy and drug exposure of a partner and refrain from donating sperm from the first administration of IMP until 3 months after the last administration of IMP. Any female partner of a non-vasectomized male patient who is of childbearing potential must use contraceptive methods with a failure rate of < 1% to prevent pregnancy (see above) from at least 2 weeks prior to the first administration of IMP to 4 weeks after the last administration of IMP.
10. Patients without contraindications for treatment with diclofenac.

Exclusion Criteria:

1. History of any clinically significant disease or disorder which, in the opinion of the Investigator, may either put the patient at risk because of participation in the trial, or influence the results or the patient's ability to participate in the trial.
2. Previous IA fracture of the knee.
3. Patient has rheumatoid arthritis, psoriatic arthritis, or has been diagnosed with any other disorders that is the primary source of their knee pain, including but not limited to: osteonecrosis, radiculopathy, bursitis, tendinitis, tumor, cancer.
4. IA injections of steroids or HA or other invasive procedure (e.g., arthroscopy, arthrography, surgery) in the knee within 3 months prior to screening.
5. Conditions or medications that could confound the assessment of pain, as judged by the Investigator.
6. Conditions that could be adversely affected by an IA injection (e.g., eczema, skin infection, high bleeding risk etc.), as judged by the Investigator.
7. Any clinically significant illness (except KOA), medical/surgical procedure, or trauma within 4 weeks of the administration of IMP.
8. Malignancy within the past 5 years, with the exception of in situ removal of basal cell carcinoma.
9. Any planned major surgery within the duration of the trial.
10. Patients who are pregnant, currently breastfeeding, or intend to become pregnant during the course of the trial.
11. Any positive result on screening for serum hepatitis B surface antigen, hepatitis C antibodies and/or human immunodeficiency virus (HIV).
12. After 10 minutes supine rest at the time of screening, any vital signs outside the following ranges:

    * Systolic blood pressure (BP): <90 or >160 mmHg, or
    * Diastolic blood pressure <50 or >95 mmHg, or
    * Pulse <40 or >90 bpm
13. Prolonged QTcF (> 450 ms), cardiac arrhythmias or any clinically significant abnormalities in the resting ECG at the time of screening, as judged by the Investigator.
14. History of severe allergy/hypersensitivity or ongoing allergy/hypersensitivity, as judged by the Investigator, or history of hypersensitivity to drugs with a similar chemical structure or class to SYN321, including disinfectants and adhesives or hypersensitivity to acetylsalicylic acid.
15. History of asthma, angioedema, urticaria or acute rhinitis induced by NSAID, including acetylsalicylic acid.
16. Regular use of any prescribed or non-prescribed medications, including but not limited to antacids, analgesics, herbal remedies, vitamins and minerals, within 10 days prior to the first administration of IMP, as well as nasal decongestants without cortisone, antihistamine, or anticholinergics for a maximum of 10 days, at the discretion of the Investigator.
17. Patient has taken pain medication or has received pain medicine other than paracetamol for conditions unrelated to KOA of the index knee within 10 days prior to the injection.
18. Planned treatment or treatment with another investigational drug within 3 months prior to Day 1. Patients consented and screened but not dosed in previous phase 1 studies will not be excluded.
19. Current smokers or users of nicotine products. Irregular use of nicotine (e.g., smoking, snuffing, chewing tobacco) less than 3 times/week before the screening visit will be allowed.
20. Positive screen for drugs of abuse or alcohol at screening. Positive results that are expected given the patient's medical history and prescribed medications can be disregarded as judged by the Investigator.
21. History of or current alcohol abuse or excessive intake of alcohol, as judged by the Investigator.
22. History of or current drug abuse, as judged by the Investigator.
23. History of or current use of anabolic steroids, as judged by the Investigator.
24. Plasma donation within 1 month of screening or blood donation (or corresponding blood loss) during the last 3 months prior to screening.
25. The Investigator considers the patient unlikely to comply with trial procedures, restrictions, and requirements.

Ages: 40 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2025-08-19 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Incidence and intensity of adverse events | From IMP injection (day 1) until end of trial visit (day 56)
  Frequency, intensity and seriousness of adverse events (AEs) will be assesed. The intensity grades is defined as mild, moderate or severe. AEs will be assessed as not related, possibly or probably related to SYN321
Clinically significant changes in ECG | From screening until end of trial visit (day 56)
  Single 12-lead ECGs will be recorded in supine position after 10 minutes of rest using an ECG machine. The resting heart rate and PQ/PR, QRS, QT and QTcF intervals will be recorded. Any values outside of normal ranges will be judged as clinically significant or not clinically significant by the Investigator. Abnormal post-IMP administration findings assessed by the Investigator as clinically significant will be reported as Adverse Events.
Clinically significant changes in blood pressure | From screening until end of trial visit (day 56)
  Systolic and diastolic blood pressure and pulse will be measured in supine positionafter 10 minutes of rest. Any vital signs outside of normal ranges will be judged as clinically significant or not clinically significant by the Investigator. Abnormal post-IMP administration findings assessed by the Investigator as clinically significant will be reported as Adverse Events.
Clinically significant changes in heart rate | From screening until end of trial visit (day 56)
  Heart rate will be measured in supine position after 10 minutes of rest. Any vital signs outside of normal ranges will be judged as clinically significant or not clinically significant by the Investigator. Abnormal post-IMP administration findings assessed by the Investigator as clinically significant will be reported as Adverse Events.
Clinically significant changes in body temperature | From screening until end of trial visit (day 56)
  Body temperature will be measured in supine position after 10 minutes of rest. Any vital signs outside of normal ranges will be judged as clinically significant or not clinically significant by the Investigator. Abnormal post-IMP administration findings assessed by the Investigator as clinically significant will be reported as Adverse Events.
Clinically significant changes in Clinical Laboratory Profile | From screening until end of trial visit (day 56)
  Safety laboratory data, Clinical chemistry, haematology, and coagulation, will be measured. Any values outside of normal ranges will be judged as clinically significant or not clinically significant by the Investigator. Abnormal post-IMP administration findings assessed by the Investigator as clinically significant will be reported as Adverse Events.
Clinically significant changes in urine analysis | From screening until end of trial visit (day 56)
  Urine analysis will be performed. Any values outside of normal ranges will be judged as clinically significant or not clinically significant by the Investigator. Abnormal post-IMP administration findings assessed by the Investigator as clinically significant will be reported as Adverse Events.
Clinically significant changes in Physical Examination | From screening until end of trial visit (day 56)
  Assessment of different organ systems. Any abnormalities will be specified and documented as clinically significant or not clinically significant. Abnormal post-IMP administration findings assessed by the Investigator as clinically significant will be reported as AEs
Clinically significant changes of local tolerability reactions | From screening until end of trial visit (day 56)
  The infusion site area will be visually inspected at baseline and follow up-visits after the IMP injection. The assessment will include the Investigator's evaluation of swelling, Redness and warmth. Abnormal post-IMP administration findings assessed by the Investigator as clinically significant will be reported as AEs.

SECONDARY OUTCOMES:
Pharmacokinetic (PK) parameter in plasma - Cmax | From IMP injection (day 1) until end of trial visit (day 56)
  Venous samples for the determination of plasma concentrations (Cmax) of diclofenac and diclofenac lactam (break down products from SYN321) will be collected.
Pharmacokinetic (PK) parameter in plasma - Cmax | From IMP injection (day 1) until end of trial visit (day 56)
  Venous samples for the determination of plasma concentrations (Cmax) of linker and linker associated metabolites (break down products from SYN321) will be collected.
Pharmacokinetic (PK) parameter in urine - Cmax | From IMP injection (day 1) until end of trial visit (day 56)
  Urine samples for the determination of plasma concentrations (Cmax) of diclofenac and diclofenac lactam (break down products from SYN321) will be collected.
Pharmacokinetic (PK) parameter in urine - Cmax | From IMP injection (day 1) until end of trial visit (day 56)
  Urine samples for the determination of plasma concentrations (Cmax) of linker and linker associated metabolites (break down products from SYN321) will be collected.
Pharmacokinetic (PK) parameter in plasma - AUC | From IMP injection (day 1) until end of trial visit (day 56)
  Venous samples for the determination of plasma concentrations (AUC) of diclofenac and diclofenac lactam (break down products from SYN321) will be collected.
Pharmacokinetic (PK) parameter in plasma - AUC | From IMP injection (day 1) until end of trial visit (day 56)
  Venous samples for the determination of plasma concentrations (AUC) of linker and linker associated metabolites (break down products from SYN321) will be collected.
Pharacokinetic (PK) parameter in urine - AUC | From IMP injection (day 1) until end of trial visit (day 56)
  Urine samples for the determination of plasma concentrations (AUC) of diclofenac and diclofenac lactam (break down products from SYN321) will be collected.
Self-registered pain in knee | From screening until end of trial visit (day 56)
  Self-registered pain using the NRS (0-10). Score 0 indicates 'no pain' and 10 indicates 'pain as bad as you can imagine'.
Self-registered function | From IMP injection until end of trial visit (day 56)
  Self-registered function using KOOS (Knee Injury and Osteoarthritis Outcome Score). Change from baseline in average sum of KOOS scores, KOOS subscale scores. The patients will assign scores (0-4, where 0 corresponds to "none" and 4 corresponds to "extreme").
Self-registered quality of life | From IMP injection until end of trial visit (day 56)
  Self-registered function using KOOS (Knee Injury and Osteoarthritis Outcome Score). Change from baseline in average sum of KOOS scores, KOOS subscale scores. The patients will assign scores (0-4, where 0 corresponds to "none" and 4 corresponds to "extreme").

CONTACTS AND LOCATIONS:
Locations (1):
- Cinical Trial Consultants AB, Uppsala, Sweden

IPD SHARING:
Plan to Share IPD: Undecided